CLINICAL TRIAL: NCT00628719
Title: A Phase III Randomized, Controlled, Clinical Trial to Assess the Safety and Efficacy of Single Infusion of Liposomal Amphotericin B in Patients With Visceral Leishmaniasis
Brief Title: Single Infusion of Liposomal Amphotericin B in Indian Visceral Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Professor Shyam Sundar, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA KAMRC
Record Dates: First submitted 2008-02-20; First posted 2008-03-05 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; India; Liposomal Amphotericin B; Amphotericin B deoxycholate
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B; amphotericin B, deoxycholate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): a single dose of 10 mg/kg of liposomal amphotericin B
  Interventions: Drug: Liposomal Amphotericin B
- 2 (Active Comparator): amphotericin B as a 1x test dose and then at a dose of 1 mg/kg/every other day for a total of 15 doses over 30 days.
  Interventions: Drug: amphotericin B deoxycholate

INTERVENTIONS:
Drug: Liposomal Amphotericin B — a single dose of 10 mg/kg of liposomal amphotericin B
  Other Names: AmBisome
  Arms: 1
Drug: amphotericin B deoxycholate — amphotericin B as a 1x test dose and then at a dose of 1 mg/kg/every other day for a total of 15 doses over 30 days.
  Arms: 2

SUMMARY:
The purpose of this trial is to evaluate the efficacy of single dose amphotericin B in the treatment of Visceral Leishmaniasis (VL) in India.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the efficacy of single dose amphotericin B in the treatment of VL in India.

Primary objective: Comparison of the efficacy of single dose of 10 mg/kg of liposomal amphotericin B to amphotericin B deoxycholate with regards to final cure rates

Secondary objective:. Comparison of the safety of single dose of 10 mg/kg of liposomal amphotericin B to amphotericin B deoxycholate when administered in the proposed dosage regimens.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults 2-65 years of age (inclusive) of either gender.
* Diagnosis of VL confirmed by spleen or bone marrow aspirate.
* Clinical signs and symptoms compatible with VL.
* Biochemical and haematological test values as follows:
* Haemoglobin > 3.5g/100mL
* White blood cell count > 0.75 x109/L
* Platelet count > 40 x 109/L
* AST, ALT and alkaline phosphatase < 5 times upper normal limit
* Prothrombin time < 4 seconds above control
* Serum creatinine levels - 1.5 times upper normal limit
* Serum potassium levels within normal limits
* HIV negative.

Exclusion Criteria:

* A history of intercurrent or concurrent diseases (e.g. chronic alcohol consumption or drug addiction; renal, hepatic, cardiovascular or CNS disease; diabetes; tuberculosis; other infectious or major psychiatric diseases) that may introduce variables that affect the outcome of the study.
* Any condition which the investigator thinks may prevent the patient from completing the study therapy and subsequent follow-up.
* Proteinuria (> 2+).
* A history of allergy or hypersensitivity to amphotericin B
* Previous treatment for VL within two weeks of enrollment into the study.
* Prior treatment failures with amphotericin B.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Final cure rate at six months after the end of treatment | One year

SECONDARY OUTCOMES:
Initial cure after the end of treatment | six months

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Study Director — Banaras Hindu University
Locations (1):
- Kala-azar Medical Research Center, Rambag Road, Muzaffarpur, India

REFERENCES:
- [Derived] Sundar S, Chakravarty J, Agarwal D, Rai M, Murray HW. Single-dose liposomal amphotericin B for visceral leishmaniasis in India. N Engl J Med. 2010 Feb 11;362(6):504-12. doi: 10.1056/NEJMoa0903627. PMID 20147716